CLINICAL TRIAL: NCT03884140
Title: Clinical Diagnostic Evaluation of Thyroid Nodules
Brief Title: Clinical Diagnostic Approach for Cases of Thyroid Nodules
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, amira hassan abd el Aziz, Assistant Lecturer, Assiut University
Other Study IDs: thyroid nodules
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Thyroid Nodule
Keywords: Thyroid nodules; T.S.H; Thyroid US; FNAC
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thyroid nodules are a common presentation in the clinic, with an increasing incidence, especially in women. Their clinical significance is mainly related to excluding malignancy (4.0 to 6.5% of all thyroid nodules).

DETAILED DESCRIPTION:
Thyroid nodule is a discrete lesion in the thyroid gland that is radiologically distinct from the surrounding thyroid parenchyma.

Thyroid nodules are a common presentation in the clinic, with an increasing incidence, especially in women. The detection rate among healthy individuals is as high as 50%-60%, but the reported incidence of malignant nodules in all thyroid nodules has ranged from only 1.6%-12%.

They are discovered either clinically on self-palpation by a patient, or during a physical examination by the clinician or incidentally during a radiologic procedure such as ultrasonography (US) imaging, computed tomography (CT) or magnetic resonance imaging (MRI) of the neck; with the increased use of sensitive imaging techniques, thyroid nodules are being diagnosed incidentally with increasing frequency in the recent years.

Though thyroid nodules are common, their clinical significance is mainly related to excluding malignancy (4.0 to 6.5% of all thyroid nodules), evaluating their functional status and if they cause pressure symptoms.

Thyroid nodules can be caused by many disorders:

Benign (colloid nodule, Hashimoto's thyroiditis, simple or hemorrhagic cyst, follicular adenoma and subacute thyroiditis) and malignant (Papillary Cancer, Follicular Cancer, Hurthle Cell Cancer, Anaplastic Cancer, Medullary Cancer, Thyroid Lymphoma and metastases).

Initial assessment of a patient found to have a thyroid nodule either clinically or incidentally should include a detailed and relevant history plus physical examination. Laboratory tests should begin with measurement of serum thyroid-stimulating hormone (TSH). Thyroid scintigraphy/radionuclide thyroid scan should be performed in patients presenting with a low serum TSH.

Thyroid ultrasound should be performed in all those suspected or known to have a nodule to confirm the presence of a nodule, evaluate for additional nodules and cervical lymph nodes and assess for suspicious sonographic features.

The next step in the evaluation of a thyroid nodule is a fine needle aspiration (FNA) biopsy, which is the gold standard diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

* all patient presented by thyroid nodules either discovered clinically or incidentally.

Exclusion Criteria:

* no

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients aged between 18-75 years presented by thyroid nodule either clinically or incidentally discovered coming to thyroid clinic for evaluation.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
correlation between clinical presentation and the results of diagnostic tools to reach to proper evaluation of thyroid nodules. | baseline
  develop a rational, cost-effective approach to ordering and interpreting imaging and diagnostic tests in the evaluation of the thyroid nodule.

REFERENCES:
- [Background] Tessler FN, Middleton WD, Grant EG, Hoang JK, Berland LL, Teefey SA, Cronan JJ, Beland MD, Desser TS, Frates MC, Hammers LW, Hamper UM, Langer JE, Reading CC, Scoutt LM, Stavros AT. ACR Thyroid Imaging, Reporting and Data System (TI-RADS): White Paper of the ACR TI-RADS Committee. J Am Coll Radiol. 2017 May;14(5):587-595. doi: 10.1016/j.jacr.2017.01.046. Epub 2017 Apr 2. PMID 28372962
- [Background] Tamhane S, Gharib H. Retraction Note: Thyroid nodules update in diagnosis and management. Clin Diabetes Endocrinol. 2016 Apr 14;2:10. doi: 10.1186/s40842-016-0025-9. eCollection 2016. PMID 28707682
- [Background] Davies L, Welch HG. Current thyroid cancer trends in the United States. JAMA Otolaryngol Head Neck Surg. 2014 Apr;140(4):317-22. doi: 10.1001/jamaoto.2014.1. PMID 24557566
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786